CLINICAL TRIAL: NCT00145119
Title: Incidence and Prediction of Life-threatening Cardiac Arrhythmias in Patients With Depressed Left Ventricular Function After Acute Myocardial Infarction
Brief Title: CARISMA : Cardiac Arrhythmias and Risk Stratification After MyoCardial Infarction
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Other Study IDs: Medtronic_BRC_CRM_001
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2018-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Cardiac arrhythmias; Left ventricular dysfunction; Implantable loop recorder; Risk stratifiers
MeSH Terms: conditions — Arrhythmias, Cardiac; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to assess the incidence of tachy- and bradyarrhythmic episodes in patients with acute myocardial infarction with depressed ventricular function and to determine the predictive value of several invasive and non-invasive risk markers for life-threatening arrhythmia

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction (< 21 days)
* Ejection fraction <= 40 % or wall motion index <= 1.3

Exclusion Criteria:

* Implantable loop recorder can't be implanted within 3 weeks after MI
* NYHA class IV
* Planned or previous ICD implantation
* Planned CABG
* Severe valvular disease
* Pregnancy
* Life expectancy < 1 year for non-cardiac cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2001-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Huikuri, Prof., Principal Investigator — Oulu University Central Hospital, Finland; P. E. Bloch-Thomsen, Dr., Principal Investigator — Gentofte University Hospital, Denmark
Locations (1):
- Medtronic Bakken Research Center B.V., Maastricht, Netherlands

REFERENCES:
- [Derived] Sakthivel T, Risum N, Bundgaard H, Joergensen RM, Jacobsen UG, Huikuri HV, Thomsen PEB, Jons C, Thomsen AF. Incidentally Induced Atrial Fibrillation During Programmed Electrical Stimulation in Patients With Depressed Left Ventricular Systolic Function After an Acute Myocardial Infarction. Ann Noninvasive Electrocardiol. 2024 Sep;29(5):e70011. doi: 10.1111/anec.70011. PMID 39225437
- [Derived] Jorgensen RM, Levitan J, Halevi Z, Puzanov N, Abildstrom SZ, Messier MD, Huikuri HV, Haarbo J, Thomsen PE, Jons C; CARISMA investigators. Heart rate variability density analysis (Dyx) for identification of appropriate implantable cardioverter defibrillator recipients among elderly patients with acute myocardial infarction and left ventricular systolic dysfunction. Europace. 2015 Dec;17(12):1848-54. doi: 10.1093/europace/euu394. Epub 2015 Mar 8. PMID 25755288
- [Derived] Ruwald AC, Gang U, Thomsen PE, Jorgensen RM, Ruwald MH, Huikuri HV, Jons C. The predictive value of CHADS(2) risk score in post myocardial infarction arrhythmias - a Cardiac Arrhythmias and RIsk Stratification after Myocardial infArction (CARISMA) substudy. Int J Cardiol. 2014 May 15;173(3):441-6. doi: 10.1016/j.ijcard.2014.03.010. Epub 2014 Mar 15. PMID 24713455
- [Derived] Ruwald AC, Bloch Thomsen PE, Gang U, Jorgensen RM, Huikuri HV, Jons C. New-onset atrial fibrillation predicts malignant arrhythmias in post-myocardial infarction patients--a Cardiac Arrhythmias and RIsk Stratification after acute Myocardial infarction (CARISMA) substudy. Am Heart J. 2013 Nov;166(5):855-63.e3. doi: 10.1016/j.ahj.2013.08.017. Epub 2013 Sep 26. PMID 24176441
- [Derived] Gang UJ, Jons C, Jorgensen RM, Abildstrom SZ, Messier MD, Haarbo J, Huikuri HV, Thomsen PE. Clinical significance of late high-degree atrioventricular block in patients with left ventricular dysfunction after an acute myocardial infarction--a Cardiac Arrhythmias and Risk Stratification After Acute Myocardial Infarction (CARISMA) substudy. Am Heart J. 2011 Sep;162(3):542-7. doi: 10.1016/j.ahj.2011.06.021. Epub 2011 Aug 11. PMID 21884874
- [Derived] Jons C, Jacobsen UG, Joergensen RM, Olsen NT, Dixen U, Johannessen A, Huikuri H, Messier M, McNitt S, Thomsen PE; Cardiac Arrhythmias and Risk Stratification after Acute Myocardial Infarction (CARISMA) Study Group. The incidence and prognostic significance of new-onset atrial fibrillation in patients with acute myocardial infarction and left ventricular systolic dysfunction: a CARISMA substudy. Heart Rhythm. 2011 Mar;8(3):342-8. doi: 10.1016/j.hrthm.2010.09.090. Epub 2010 Nov 18. PMID 21093611
- [Derived] Bloch Thomsen PE, Jons C, Raatikainen MJ, Moerch Joergensen R, Hartikainen J, Virtanen V, Boland J, Anttonen O, Gang UJ, Hoest N, Boersma LV, Platou ES, Becker D, Messier MD, Huikuri HV; Cardiac Arrhythmias and Risk Stratification After Acute Myocardial Infarction (CARISMA) Study Group. Long-term recording of cardiac arrhythmias with an implantable cardiac monitor in patients with reduced ejection fraction after acute myocardial infarction: the Cardiac Arrhythmias and Risk Stratification After Acute Myocardial Infarction (CARISMA) study. Circulation. 2010 Sep 28;122(13):1258-64. doi: 10.1161/CIRCULATIONAHA.109.902148. Epub 2010 Sep 13. PMID 20837897
- [Derived] Gang UJ, Jons C, Jorgensen RM, Abildstrom SZ, Haarbo J, Messier MD, Huikuri HV, Thomsen PE; CARISMA investigators. Heart rhythm at the time of death documented by an implantable loop recorder. Europace. 2010 Feb;12(2):254-60. doi: 10.1093/europace/eup383. Epub 2009 Dec 16. PMID 20019013
- [Derived] Huikuri HV, Raatikainen MJ, Moerch-Joergensen R, Hartikainen J, Virtanen V, Boland J, Anttonen O, Hoest N, Boersma LV, Platou ES, Messier MD, Bloch-Thomsen PE; Cardiac Arrhythmias and Risk Stratification after Acute Myocardial Infarction study group. Prediction of fatal or near-fatal cardiac arrhythmia events in patients with depressed left ventricular function after an acute myocardial infarction. Eur Heart J. 2009 Mar;30(6):689-98. doi: 10.1093/eurheartj/ehn537. Epub 2009 Jan 20. PMID 19155249

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients
Started | 312
Completed | 267
Not Completed | 45
Not completed — Death | 45

BASELINE CHARACTERISTICS:
Population: Survivors of an acute Myocardial Infarction (AMI) with impaired left ventricular ejection fraction
Groups:
- Patients: Survivors of an acute Myocardial Infarction (AMI) with impaired left ventricular ejection fraction
Arm/Group | Patients
Number analyzed (Participants) | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 239
Diabetes [Number; unit: participants] | 62
Ejection fraction index < 7 days after index MI [Mean (Standard Deviation); unit: percent] | 31 (6)
Pior MI [Number; unit: participants] | 116

OUTCOME MEASURES:

1. Primary Outcome: ECG-documented Ventricular Fibrillation or Symptomatic Sustained Ventricular Tachycardia (VT)
Description: ECG-documented ventricular fibrillation or symptomatic sustained ventricular tachycardia (VT)
Time Frame: 2 year
Measure: Number; unit: participants
Arm/Group | Patients
Number analyzed (Participants) | 312
participants
  Primary endoints | 25
  Sudden death | 8
  Resuscitated cardiac arrest | 3
  Syncope | 2
  Symptomatic sustained VT | 12
Statistical Analysis 1: Comparison: Patients; Test type: Superiority or Other; proportion (%) = 8

ADVERSE EVENTS:
Time Frame: Other (non-serious) adverse events were not collected/ assessed
Description: Other (non-serious) adverse events were not collected/ assessed
Arm/Group | Patients
Serious Adverse Events (participants affected / at risk) | 38/312
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=312)
Death (Cardiac disorders) | 38 (38) — Cardiac death.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No